CLINICAL TRIAL: NCT05034406
Title: The Effect of Subcutaneous and Intraperitoneal Instillation of Local Anesthetics on Postoperative Pain After Laparoscopic Varicocelectomy: A Randomized Controlled Trial
Brief Title: The Effect of Subcutaneous and Intraperitoneal Anesthesia on Post Laparoscopic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KBC Split (Other)
Responsible Party: Principal Investigator, Goran Tintor, Medical doctor, surgery resident, KBC Split
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 500-03/20-01/09
Record Dates: First submitted 2021-08-09; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Varicocele; Postoperative Pain
MeSH Terms: conditions — Varicocele; Pain, Postoperative | interventions — Lidocaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine group (Experimental): A total amount of 6 mL of 2% lidocaine was injected at the three trocar insertion sites (2 mL at each insertion site) prior to incision and 10 mL of 2% lidocaine was injected at the end of procedure, under the direct visualization of laparoscope, below and around the defect of the peritoneum at the site of varicocele.
  Interventions: Drug: 2% Lidocaine
- Levobupivacaine (Experimental): Total amount of 6 mL of 0.5% levobupivacaine was injected at the three trocar insertion sites (2 mL at each) prior to incision and 10 mL of 2% lidocaine was injected at the end of procedure, under the direct visualization of laparoscope, below and around the defect of the peritoneum at the site of varicocele.
  Interventions: Drug: 0.5% levobupivacaine
- Control group (No Intervention): No local or peritoneal administration of any local anesthetic prior, during and after the surgical procedure

INTERVENTIONS:
Drug: 2% Lidocaine — 6 mL of 2% lidocaine injected at the trocar insertion site.
  Arms: Lidocaine group
Drug: 0.5% levobupivacaine — 6 mL of 0.5% levobupivacaine injected at the trocar insertion site.
  Arms: Levobupivacaine

SUMMARY:
Aim of this study is to examine the effects of subcutaneously applied local anesthetics at trocar site in combination with intraoperative intraperitoneal analgesia on duration and character of pain in pediatric patients undergoing laparoscopic varicocelectomy.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients with varicocele who underwent laparoscopic varicocelectomy
* pediatric patients whose parents or guardians gave informed consent

Exclusion Criteria:

* patients who received open or microsurgical varicocelectomy
* pediatric patients who underwent conversion to open procedure
* pediatric patients with chronic, metabolic and endocrine diseases
* pediatric patients with systemic infections

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Pain (as measured by Visual analogue scale) | 6 hours after surgery
  Visual analogue scale (VAS, 0-10 scale with 10 being the strongest pain) of pain assessed by a blinded investigator.

SECONDARY OUTCOMES:
Pain (as measured by Visual analogue scale) | 2 hours after surgery
  Visual analogue scale (VAS, 0-10 scale with 10 being the strongest pain) of pain assessed by a blinded investigator.
Pain (as measured by Visual analogue scale) | 12 hours after surgery
  Visual analogue scale (VAS, 0-10 scale with 10 being the strongest pain) of pain assessed by a blinded investigator.
Pain (as measured by Visual analogue scale) | 24 hours after surgery
  Visual analogue scale (VAS, 0-10 scale with 10 being the strongest pain) of pain assessed by a blinded investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Zenon Pogorelić, MD, PhD, Study Chair — University of Split, School of Medicine
Locations (1):
- University Hospital Split, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: No